CLINICAL TRIAL: NCT04519645
Title: A Multicenter, Open-Label, Randomized, Active Comparator Study to Evaluate the Efficacy, Safety, and Pharmacokinetics of Lacosamide in Neonates With Repeated Electroencephalographic Neonatal Seizures
Brief Title: A Study to Evaluate the Efficacy, Safety, and Pharmacokinetics of Lacosamide in Neonates With Repeated Electroencephalographic Neonatal Seizures
Acronym: LENS
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Study stopped after agreed PIP modification, not linked to safety reasons.
Sponsor: UCB Biopharma SRL (Industry)
Responsible Party: Sponsor
Organization: UCB Pharma (Industry)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: SP0968; 2020-001066-10 (EudraCT Number)
Record Dates: First submitted 2020-07-31; First posted 2020-08-20 (Actual); Results first posted 2025-10-03 (Actual); Last update posted 2025-10-03 (Actual); Status verified 2025-09

CONDITIONS: Electroencephalographic Neonatal Seizures; Epilepsy
Keywords: electroencephalographic neonatal seizures; epilepsy; neonatal study participants; Vimpat; lacosamide; LCM; pediatric; video-EEG
MeSH Terms: conditions — Epilepsy | interventions — Lacosamide

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- Lacosamide (Experimental): Study participants randomized to this arm will receive lacosamide (LCM) as an intravenous infusion in the Treatment Period and may continue to receive lacosamide in the Extension Period. Participants should be switched to oral dosing of LCM as soon as medically possible during the Extension Period.
  Interventions: Drug: Lacosamide intravenous; Drug: Lacosamide oral
- Active Comparator (Active Comparator): Study participants randomized to this arm will receive Active Comparator chosen based on standard of care (StOC) in the Clinical Practice in the Treatment Period and may continue to receive in the Extension Period.
  Interventions: Other: Active Comparator

INTERVENTIONS:
Drug: Lacosamide intravenous — Study participants will receive lacosamide (LCM) as an intravenous (iv) infusion during the Treatment Period.
  Other Names: LCM
  Arms: Lacosamide
Drug: Lacosamide oral — Study participants may receive lacosamide (LCM) as an oral solution during the Extension Period.
  Other Names: LCM
  Arms: Lacosamide
Other: Active Comparator — Active Comparator treatment will be chosen and dosed based on StOC (per local practice and treatment guidelines).
  Arms: Active Comparator

SUMMARY:
The purpose of the study is to evaluate the efficacy of lacosamide (LCM) versus an Active Comparator chosen based on standard of care (StOC) in severe and nonsevere seizure burden (defined as total minutes of electroencephalographic neonatal seizures (ENS) per hour) in neonates with seizures that are not adequately controlled with previous anti-epileptic drug (AED) treatment.

ELIGIBILITY:
Inclusion Criteria:

* Participant must be ≥34 weeks of corrected gestational age (CGA), <46 weeks of CGA, and <28 days of postnatal age (PNA)
* Participants who have confirmation on video-electroencephalogram (EEG) of ≥2 minutes of cumulative electroencephalographic neonatal seizures (ENS) or ≥3 identifiable ENS prior to entering the Treatment Period
* Participants must have received either phenobarbital (PB), levetiracetam (LEV), or midazolam (MDZ) (in any combination) before entering the study
* Participant weighs at least 2.3 kg at the time of enrollment Informed consent
* An Independent Ethics Committee (IEC)-approved written informed consent form (ICF) is signed and dated by the participant's parent(s) or legal representative(s)

Exclusion Criteria:

* Participant with seizures responding to correction of metabolic disturbances (hypoglycemia, hypomagnesemia, or hypocalcemia) or with seizures for which a targeted, known treatment is available
* Participant has seizures related to prenatal maternal drug use or drug withdrawal
* Participant has a clinically relevant electrocardiogram (ECG) abnormality, in the opinion of the investigator
* Participant receiving treatment with phenytoin (PHT), lidocaine (LDC), or other sodium channel blockers at any time

Max Age: 28 Days | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 29 (Actual)
Dates: Start 2021-03-31 (Actual); Primary Completion 2024-08-06 (Actual); Study Completion 2024-10-31 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: UCB Cares, Study Director — 001 844 599 2273
Locations (18):
- United States (15):
  - Sp0968 101, La Jolla, California
  - Sp0968 108, Long Beach, California
  - Sp0968 116, Los Angeles, California
  - Sp0968 190, San Diego, California
  - Sp0968 118, Aurora, Colorado
  - Sp0968 104, Jacksonville, Florida
  - Sp0968 107, Miami, Florida
  - Sp0968 112, Iowa City, Iowa
  - Sp0968 125, Valhalla, New York
  - Sp0968 117, Portland, Oregon
  - Sp0968 109, Austin, Texas
  - Sp0968 192, Salt Lake City, Utah
  - Sp0968 105, Salt Lake City, Utah
  - Sp0968 102, Charlottesville, Virginia
  - Sp0968 122, Seattle, Washington
- Australia (2):
  - Sp0968 302, Parkville
  - Sp0968 301, South Brisbane
- Sp0968 201, Toronto, Canada

IPD SHARING:
Plan to Share IPD: Yes
Data from this trial may be requested by qualified researchers six months after product approval in the US and/or Europe, or global development is discontinued, and 18 months after trial completion. Investigators may request access to anonymized individual patient-level data and redacted trial documents which may include: analysis-ready datasets, study protocol, annotated case report form, statistical analysis plan, dataset specifications, and clinical study report. Prior to use of the data, proposals need to be approved by an independent review panel at www.Vivli.org and a signed data sharing agreement will need to be executed. All documents are available in English only, for a prespecified time, typically 12 months, on a password protected portal. This plan may change if the risk of re-identifying trial participants is determined to be too high after the trial is completed; in this case and to protect participants, individual patient-level data would not be made available.
Supporting Information: Study Protocol, SAP, CSR
Time Frame: Data from this trial may be requested by qualified researchers six months after product approval in the US and/or Europe or global development is discontinued, and 18 months after trial completion.
Access Criteria: Qualified researchers may request access to anonymized IPD and redacted study documents which may include: raw datasets, analysis-ready datasets, study protocol, blank case report form, annotated case report form, statistical analysis plan, dataset specifications, and clinical study report. Prior to use of the data, proposals need to be approved by an independent review panel at www.Vivli.org and a signed data sharing agreement will need to be executed.All documents are available in English only, for a pre-specified time, typically 12 months, on a password protected portal.
URL: https://www.Vivli.org

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The study started to enrol participants in March 2021 and concluded in October 2024.
Pre-assignment Details: The Participant Flow refers to the Safety set. This study was ended after agreed Pediatric investigation plan (PIP) modification, not linked to safety reasons.
Groups:
- No Treatment: Participant signed the informed consent form, successfully screened and randomized but never received any study medication during the study.
- Active Comparator: Study participants randomized to receive Active Comparator (chosen and dosed based on standard of care (StOC) per local practice and treatment guidelines) in the Treatment Period. After the Treatment Period, study participants had the option to continue to receive randomized Active Comparator in the Extension Period (up to 28 days of postnatal age). Study participants (whether they discontinued randomized treatment during the Treatment Period, completed the Extension Period, were discharged from the hospital, or reached 28 days of postnatal age) then entered the 14-day Safety Follow-up (SFU) Period with optional down titration.
- Lacosamide: Study participants randomized to receive lacosamide 10 milligram per milliliter (mg/mL) 3 times a day as an intravenous infusion over 30 minutes for up to 96 hours in the Treatment Period. After the Treatment Period, study participants had the option to continue to receive randomized lacosamide in the Extension Period (up to 28 days of postnatal age), being switched to oral dosing of lacosamide as soon as medically possible. Study participants (whether they discontinued randomized treatment during the Treatment Period, completed the Extension Period, were discharged from the hospital, or reached 28 days of postnatal age) then entered the 14-day SFU Period with optional down titration.
Period: Enrollment Period (Up to 36 Hours)
Arm/Group | No Treatment | Active Comparator | Lacosamide
Started | 3 | 11 | 15
Completed | 0 | 11 | 15
Not Completed | 3 | 0 | 0
Not completed — Adverse Event | 1 | 0 | 0
Not completed — Withdrawal by Parent/Guardian | 1 | 0 | 0
Not completed — Protocol Violation | 1 | 0 | 0
Period: Treatment Period (Up to 96 Hours)
Arm/Group | No Treatment | Active Comparator | Lacosamide
Started ((Randomized)) | 0 | 11 | 15
Safety Set (Actual Treated) | 0 | 12 (One participant was randomized to lacosamide but received active comparator. Thus, one additional participant is included in the active comparator population for safety analyses.) | 14
Full Analysis Set (Treated as Randomized) | 0 | 9 | 15
Completed | 0 | 10 | 15
Not Completed | 0 | 1 | 0
Not completed — Consent withdrawn by parent/guardian,not due to AE | 0 | 1 | 0
Period: Extension Period: up to 28 Days of PNA
Arm/Group | No Treatment | Active Comparator | Lacosamide
Started | 0 | 0 (No participant taking Active Comparator opted to continue in the Extension Period.) | 12 (Out of 15 randomized participants who completed the Treatment Period, 12 participants opted to continue in the Extension Period.)
Completed | 0 | 0 | 12
Not Completed | 0 | 0 | 0
Period: Safety Follow Up Period: 14 Days
Arm/Group | No Treatment | Active Comparator | Lacosamide
Started | 0 | 10 (All of the study participants who completed the Treatment Period entered the Safety Follow-up Period. The one participant in the Active Comparator arm, who did not complete the treatment period, did not enter the Safety Follow-up Period.) | 15 (All of the study participants (including those who completed the Extension Period and the three participants who did not opt to continue in the Extension Period) entered the Safety Follow-up Period.)
Completed | 0 | 10 | 15
Not Completed | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Population: The Safety Set (SS) consisted of all enrolled study participants who took at least 1 dose of the randomized treatment. The safety population was based on actual treatment. As pre-defined in the SAP, Baseline data was collected and reported for Treated population only.
Groups:
- Total: Total of all reporting groups
Arm/Group | Active Comparator | Lacosamide | Total
Number analyzed (Participants) | 12 | 14 | 26
Age, Continuous [Mean (Standard Deviation); unit: days] | 3.1 (2.8) | 4.1 (5.0) | 3.7 (4.1)
Age, Customized [Count of Participants; unit: Participants]
  0-<=27 days | 12 | 14 | 26
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 7 | 7 | 14
  Male | 5 | 7 | 12
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 4 | 7 | 11
  Not Hispanic or Latino | 7 | 6 | 13
  Unknown or Not Reported | 1 | 1 | 2
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Race: Black or African American | 1 | 0 | 1
  Race: White | 8 | 11 | 19
  Race: Other or Mixed | 2 | 2 | 4
  Race: Missing | 1 | 1 | 2

OUTCOME MEASURES:

1. Primary Outcome: Change in Seizure Burden Measured in the Evaluation Video-electroencephalogram (Video-EEG) Compared With the Baseline Video-EEG
Description: Baseline seizure burden was defined as seizure burden measured on the continuous video-EEG (total electroencephalographic neonatal seizures (ENS) in minutes per hour) during a period of up to 2 hours immediately prior to the first administration of study drug. An ENS was defined as an EEG seizure lasting for at least 10 seconds on video-EEG. The seizure burden in the Evaluation Period was calculated as the total duration of seizures between 1 and 3 hours after the first dose of study medication divided by the duration of interpretable video-EEG available in the same period. Change in seizure burden measured in the Evaluation video-EEG compared with the Baseline video-EEG was analyzed such that a positive value indicates a reduction in seizure burden from baseline.
Time Frame: During 2-hour Evaluation starting 1 hour after initial treatment (up to 2 hours), compared to Baseline
Population: The Full Analysis Set (FAS) consisted of all study participants in the SS who had a minimum of 30 minutes of interpretable video-EEG data from both Baseline and the period between 1 and 3 hours (Evaluation Period) after randomization to the initial study medication treatment. The FAS population was based on randomized treatment. Here, overall number of participants analyzed included all participants who were evaluable for this assessment.
Measure: Mean (Standard Deviation); unit: minute per hour (min/hour)
Arm/Group | Active Comparator | Lacosamide
Number analyzed (Participants) | 9 | 11
minute per hour (min/hour) | 2.45 (14.83) | 6.64 (6.55)

2. Secondary Outcome: Percentage of Responders in the Evaluation Video-EEG Compared With the Baseline Video-EEG
Description: A responder is defined as a study participant who achieved the following reduction in seizure burden without need for rescue medication, compared with the seizure burden measured during the Baseline Period immediately prior to the study medication administration, evaluated for a 2-hour period starting 1 hour after the start of initial treatment: - At least 80% reduction of seizure burden in participants who were categorized by the Investigator as having non-severe seizure burden during Baseline OR - At least 50% reduction of seizure burden in participants who were categorized by the Investigator as having severe seizure burden during Baseline.
Time Frame: During 2-hour Evaluation starting 1 hour after initial treatment (up to 2 hours), compared to Baseline
Population: The FAS consisted of all study participants in the SS who had a minimum of 30 minutes of interpretable video-EEG data from both Baseline and the period between 1 and 3 hours (Evaluation Period) after randomization to the initial study medication treatment. The FAS population was based on randomized treatment.
Measure: Number; unit: percentage of participants
Arm/Group | Active Comparator | Lacosamide
Number analyzed (Participants) | 9 | 15
percentage of participants | 66.7 | 60.0

3. Secondary Outcome: Percentage of Participants With at Least 80% Reduction in Seizure Burden in the Evaluation a Video-EEG Compared With the Baseline Video-EEG
Description: A responder is defined as a study participant who achieved the following reduction in seizure burden without need for rescue medication, compared with the seizure burden measured during the Baseline Period immediately prior to investigational medicinal product (IMP) administration, evaluated for a 2-hour period starting 1 hour after the start of initial treatment: A reduction in seizure burden from Baseline of >=80% regardless of baseline seizure severity. Percentage of Participants With at least 80% Reduction in Seizure Burden in the Evaluation (starting 1 hour after treatment) of a Video-EEG Compared with the Baseline Video-EEG were reported.
Time Frame: During 2-hour Evaluation starting 1 hour after initial treatment (up to 2 hours), compared to Baseline
Population: as for outcome 2
Measure: Number; unit: percentage of participants
Arm/Group | Active Comparator | Lacosamide
Number analyzed (Participants) | 9 | 15
percentage of participants | 44.4 | 60.0

4. Secondary Outcome: Time to Response Across the 48-hour Treatment Period Compared With the Baseline Video-EEG
Description: Time to response where response was defined as a reduction in seizure burden from Baseline of at least 80% in participants with non-severe seizure burden, and of at least 50% for participants with severe seizure burden. Time to response was censored at the date/time the participant received rescue medication or stopped video-EEG monitoring, or otherwise at the end of the 48-hour period.
Time Frame: Across the first 48 hours of Treatment Period, compared to Baseline
Population: as for outcome 2
Measure: Median (95% Confidence Interval); unit: hours
Arm/Group | Active Comparator | Lacosamide
Number analyzed (Participants) | 9 | 15
hours | 3.0 [3.0 to 8.0] | 3.0 [NA to NA] — Upper and lower limits of 95% confidence interval could not be calculated by the Kaplan-Meier model due to heavy censoring occurring before the median survival time was observed and a lack of variability in the response times (9/10 patients reported the same time to response).

5. Secondary Outcome: Time to Seizure Freedom Across the First 48-hour Treatment Period Compared With the Baseline Video-EEG
Description: Seizure freedom was defined as 0 minutes of seizures in a 1-hour period (or 2-hour period for the 3-hour time point) and was analyzed across the 48 hours. The time to seizure freedom was measured in hours, defined as the first time point when the response criterion was met minus the date and time of the first dose of randomized study medication administration. Time to seizure freedom was censored at the time of receiving rescue medication, stopping video-EEG monitoring or otherwise at 48 hours after first dose.
Time Frame: Across the first 48 hours of Treatment Period, compared to Baseline
Population: as for outcome 2
Measure: Median (95% Confidence Interval); unit: hours
Arm/Group | Active Comparator | Lacosamide
Number analyzed (Participants) | 9 | 15
hours | 8.0 [3.0 to NA] — Upper limit of 95% confidence interval could not be calculated by the Kaplan-Meier model due to heavy censoring occurring before the median survival time was observed and a lack of variability in the response times (4/6 patients reported the same time to seizure freedom). | 3.0 [NA to NA] — Upper and lower limits of 95% confidence interval could not be calculated by the Kaplan-Meier model due to heavy censoring occurring before the median survival time was observed and a lack of variability in the response times (9/10 patients reported the same time to seizure freedom).

6. Secondary Outcome: Absolute Change in Seizure Burden Across the First 48-hours of the Treatment Period Measured by Continuous Video-EEG Compared With the Baseline Video-EEG
Description: Baseline seizure burden was calculated as total duration of seizures (in minutes) between -2 hour and 0 hours before first dose of study medication divided by total duration of interpretable video-EEG (in hours) in the same period. Seizure burden for 8, 16, 24, 32, 40 and 48 hour time points was calculated as total duration of seizures in the hour prior to time point divided by duration of interpretable video-EEG available in same period. If <30 minutes of interpretable video-EEG were available in the 1 hour prior to the time point, response was calculated based on seizure burden for most recent 30 minutes of interpretable video-EEG in the 2 hours (for 8 and 16 hour points) or 4 hours (for 24, 32, 40 and 48 hour points) prior to time point. The 30 minutes of video-EEG did not need to be continuous. Absolute reduction in seizure burden for these time points was calculated as seizure burden in Baseline Period minus seizure burden at that time point.
Time Frame: Treatment Period: 7-8 hours, 15-16 hours, 23-24 hours, 31-32 hours, 39-40 hours, 47-48 hours, compared to Baseline
Population: FAS consisted of all study participants in the SS who had a minimum of 30 minutes of interpretable video-EEG data from both Baseline and the period between 1 and 3 hours (Evaluation Period) after randomization to the initial study medication treatment. FAS population was based on randomized treatment. Here, overall number of participants analyzed included all participants who were evaluable for this assessment and number analyzed signifies participants who were evaluable at specified timepoints.
Measure: Mean (Standard Deviation); unit: mins/hour
Arm/Group | Active Comparator | Lacosamide
Number analyzed (Participants) | 6 | 11
mins/hour
  Treatment, 7 hour - 8 hour | -2.74 (15.53) | 6.30 (6.74)
  Treatment, 15 hour - 16 hour: number analyzed (Participants) | 6 | 10
  Treatment, 15 hour - 16 hour | 3.63 (5.28) | 7.21 (6.33)
  Treatment, 23 hour - 24 hour: number analyzed (Participants) | 6 | 10
  Treatment, 23 hour - 24 hour | 5.08 (4.81) | 8.69 (8.06)
  Treatment, 31 hour - 32 hour: number analyzed (Participants) | 5 | 10
  Treatment, 31 hour - 32 hour | 5.71 (5.09) | 8.93 (8.56)
  Treatment, 39 hour - 40 hour: number analyzed (Participants) | 4 | 10
  Treatment, 39 hour - 40 hour | 4.43 (5.80) | 8.93 (8.56)
  Treatment, 47 hour - 48 hour: number analyzed (Participants) | 4 | 10
  Treatment, 47 hour - 48 hour | 4.84 (5.44) | 8.93 (8.56)

7. Secondary Outcome: Percent Change in Seizure Burden Across the First 48-hours of the Treatment Period Measured by Continuous Video-EEG Compared With the Baseline Video-EEG
Description: The percent change in seizure burden for the 8, 16, 24, 32, 40 and 48 hour time points was calculated as the seizure burden at Baseline minus the seizure burden at the respective time point, divided by the seizure burden in the Baseline Period, multiplied by 100. Percent change in seizure burden was analyzed such that a positive value indicates a reduction in seizure burden from baseline.
Time Frame: Treatment Period: 7-8 hours, 15-16 hours, 23-24 hours, 31-32 hours, 39-40 hours, 47-48 hours, compared to Baseline
Population: as for outcome 6
Measure: Mean (Standard Deviation); unit: percent change
Arm/Group | Active Comparator | Lacosamide
Number analyzed (Participants) | 6 | 11
percent change
  Treatment, 7 hour - 8 hour | 39.85 (147.33) | 80.92 (45.56)
  Treatment, 15 hour - 16 hour: number analyzed (Participants) | 6 | 10
  Treatment, 15 hour - 16 hour | 48.22 (116.94) | 93.19 (21.53)
  Treatment, 23 hour - 24 hour: number analyzed (Participants) | 6 | 10
  Treatment, 23 hour - 24 hour | 100.00 (0.00) | 99.03 (3.05)
  Treatment, 31 hour - 32 hour: number analyzed (Participants) | 5 | 10
  Treatment, 31 hour - 32 hour | 100.00 (0.00) | 100.00 (0.00)
  Treatment, 39 hour - 40 hour: number analyzed (Participants) | 4 | 10
  Treatment, 39 hour - 40 hour | 77.13 (45.73) | 100.00 (0.00)
  Treatment, 47 hour - 48 hour: number analyzed (Participants) | 4 | 10
  Treatment, 47 hour - 48 hour | 100.00 (0.00) | 100.00 (0.00)

8. Secondary Outcome: Percentage of Responders at the End of the First 48-hours of the Treatment Period
Description: A responder is defined as a study participant who achieved the following reduction in seizure burden without need for rescue medication, compared with the seizure burden measured during the Baseline Period immediately prior to investigational medicinal product (IMP) administration, evaluated for a 2-hour period starting 1 hour after the start of initial treatment: At least 80% reduction of seizure burden in participants who were categorized as having nonsevere seizure burden during Baseline OR At least 50% reduction of seizure burden in participants who had at least one 30-minute period of severe seizure burden during Baseline. The denominator for the percentages was based on the number of participants with video- EEG data available at the 48 hour time point.
Time Frame: Across the first 48 hours of Treatment Period
Population: The FAS consisted of all study participants in the SS who had a minimum of 30 minutes of interpretable video-EEG data from both Baseline and the period between 1 and 3 hours (Evaluation Period) after randomization to the initial study medication treatment. FAS population was based on randomized treatment. Here, overall number of participants analyzed included all participants who were evaluable for this assessment.
Measure: Number; unit: percentage of participants
Arm/Group | Active Comparator | Lacosamide
Number analyzed (Participants) | 6 | 13
percentage of participants | 66.7 | 76.9

9. Secondary Outcome: Percentage of Study Participants Who Are Seizure-free (100% Reduction in Seizure Burden From Baseline) at 24 Hours After Start of the Treatment Period, Categorized by Study Participants With Non Severe or Severe Seizure Burden at Baseline
Description: Seizure free was defined as 100% reduction in seizure burden or having no seizures in the assessment period (23 to 24 hours after first dose) from Baseline. For the study participants with severe seizure burden at Baseline (as determined by the Investigator), the numerator was defined as the number of participants with severe seizure burden at Baseline who had no seizures between 23 and 24 hours after the start of the Treatment Period. The denominator for the percentages was based on the number of participants with video-EEG data available at the 24 hour time point. Here, N='overall number of participants analyzed' and n='number analyzed' in categories.
Time Frame: 24 hours after the start of Treatment Period, compared to Baseline
Population: FAS consisted of all study participants in the SS who had minimum of 30 minutes of interpretable video-EEG data from both Baseline and period between 1 and 3 hours (Evaluation Period) after randomization to initial study medication treatment. FAS population was based on randomized treatment. Here, "N"=participants who were evaluable for this assessment and "n"= participants who were evaluable for specified seizure burden categories.
Measure: Number; unit: percentage of participants
Arm/Group | Active Comparator | Lacosamide
Number analyzed (Participants) | 8 | 14
percentage of participants
  Severe Seizure Burden: number analyzed (Participants) | 3 | 6
  Severe Seizure Burden | 33.3 | 66.7
  Non-severe Seizure Burden: number analyzed (Participants) | 5 | 8
  Non-severe Seizure Burden | 100.0 | 62.5

10. Secondary Outcome: Categorized Percentage of Participants With Change in Seizure Burden in the Evaluation Video-EEG Compared With the Baseline Video-EEG
Description: Baseline seizure burden was calculated as total duration of seizures (in minutes) between -2 and 0 hours before the first dose of study medication divided by total duration of interpretable video-EEG (in hours) in same period. Seizure burden in Evaluation Period was calculated as total duration of seizures between 1 and 3 hours after first dose of study medication divided by duration of interpretable video-EEG available in same period. Percent change in seizure burden for Evaluation period was calculated as seizure burden at Baseline minus seizure burden at respective time point, divided by seizure burden in Baseline Period, multiplied by 100. Participants classified in one of following categories based on their percent reduction from Baseline to Evaluation Period: < -25% (worsening), -25% to <25% (no change), 25% to <50%, 50% to <80%, and >=80%. Percent change in seizure burden was analyzed and categorized such that positive value indicates reduction in seizure burden from baseline.
Time Frame: During 2-hour Evaluation starting 1 hour after initial treatment (up to 2 hours), compared to Baseline
Population: FAS consisted of all study participants in the SS who had minimum of 30 minutes of interpretable video-EEG data from both Baseline and period between 1 and 3 hours (Evaluation Period) after randomization to the initial study medication treatment. FAS population was based on randomized treatment. Here, overall number of participants analyzed included all participants who were evaluable for this assessment.
Measure: Number; unit: Percentage of participants
Arm/Group | Active Comparator | Lacosamide
Number analyzed (Participants) | 9 | 11
Percentage of participants
  Evaluation, 1 hour - 3 hour: <-25% | 22.2 | 0.0
  Evaluation, 1 hour - 3 hour: -25% to <25% | 0.0 | 9.1
  Evaluation, 1 hour - 3 hour: 25% to <50% | 11.1 | 9.1
  Evaluation, 1 hour - 3 hour: 50% to <80% | 22.2 | 0.0
  Evaluation, 1 hour - 3 hour: >=80% | 44.4 | 81.8

11. Secondary Outcome: Percentage of Participants With Treatment-emergent Adverse Events (TEAEs) as Reported by the Investigator
Description: An adverse event (AE) is any untoward medical occurrence in a patient or clinical study participant, temporally associated with the use of study medication, whether or not considered related to the study medication. TEAEs are defined as AEs which have onset on or after the start date and time of initial study medication administration.
Time Frame: From first administration of study treatment to the End of Safety Follow-up Period (up to Day 42)
Population: The SS consisted of all enrolled study participants who took at least 1 dose of the randomized treatment. The safety population was based on actual treatment.
Measure: Number; unit: percentage of participants
Arm/Group | Active Comparator | Lacosamide
Number analyzed (Participants) | 12 | 14
percentage of participants | 41.7 | 64.3

12. Secondary Outcome: Percentage of Participants With Treatment-emergent Marked Abnormalities in 12-lead Electrocardiogram (ECG)
Description: The ECG treatment-emergent marked abnormalities values are based on grade 2 toxicity based on abnormal values or clinical experience based on investigator's discretion. Participants randomized to Lacosamide and enrolled under this version of the protocol have planned assessments at Screening, 1-6 hours, 48, and 96 hours only. For participants randomized to Active Comparator treatment, only the Screening assessment was applicable.
Time Frame: Active Comparator: Screening; Lacosamide: Screening, 1-6 hours, 48 and 96 hours
Population: The SS consisted of all enrolled study participants who took at least 1 dose of the randomized treatment. The safety population was based on actual treatment. Here, overall number of participants analyzed included all participants with a non-missing interpretation for this assessment and number analyzed signifies participants who were evaluable at specified timepoints.
Measure: Number; unit: percentage of participants
Arm/Group | Active Comparator | Lacosamide
Number analyzed (Participants) | 8 | 14
percentage of participants
  Screening: Abnormal Clinically significant | 0.0 | 0.0
  1-6 hours: Abnormal Clinically significant: number analyzed (Participants) | 0 | 9
  1-6 hours: Abnormal Clinically significant |  | 0.0
  48 hours: Abnormal Clinically significant: number analyzed (Participants) | 0 | 13
  48 hours: Abnormal Clinically significant |  | 0.0
  96 hours: Abnormal Clinically significant: number analyzed (Participants) | 0 | 12
  96 hours: Abnormal Clinically significant |  | 0.0

13. Secondary Outcome: Serum Concentration of Lacosamide
Description: Serum concentrations of lacosamide were measured and concentration data were summarized. PK sparse sampling was performed.
Time Frame: Day 1: 30-90 minutes and 6 - 8 hours after start of first infusion, 30 - 90 minutes and 6 - 8 hours after start of second or third infusion, Days 2, 3 and 4
Population: The Pharmacokinetic Per-Protocol Set (PK-PPS) consisted of all study participants who provide at least 1 measurable serum sample (with recorded sampling time) on at least 1 post-Baseline visit with documented study drug intake times. Here, overall number of participants analyzed included all participants who were evaluable for this assessment and number analyzed signifies participants who were evaluable at specified timepoints.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: microgram per milliliter (mcg/mL)
Arm/Group | Lacosamide
Number analyzed (Participants) | 13
microgram per milliliter (mcg/mL)
  Day 1: 30 - 90 minutes after start of first infusion: number analyzed (Participants) | 11
  Day 1: 30 - 90 minutes after start of first infusion | 7.003 (37.6)
  Day 1: 6 - 8 hours after start of first infusion: number analyzed (Participants) | 12
  Day 1: 6 - 8 hours after start of first infusion | 5.949 (38.6)
  Day 1: 30 - 90 minutes after start of second or third infusion: number analyzed (Participants) | 11
  Day 1: 30 - 90 minutes after start of second or third infusion | 13.27 (29.4)
  Day 1: 6 - 8 hours after start of second or third infusion | 9.607 (39.8)
  Day 2: number analyzed (Participants) | 1
  Day 2 | NA (NA) — Geometric mean and Geometric Coefficient of Variation could not be calculated for a single participant.
  Day 3: number analyzed (Participants) | 2
  Day 3 | NA (NA) — Geometric mean and Geometric Coefficient of Variation could not be calculated for less than 3 participants.
  Day 4: number analyzed (Participants) | 2
  Day 4 | NA (NA) — Geometric mean and Geometric Coefficient of Variation could not be calculated for less than 3 participants.

ADVERSE EVENTS:
Time Frame: Enrolment: Screening (-36 hours) up to 0 hours (pre-dose); Treatment: From first administration of study treatment to the End of Safety Follow-up (up to Day 42)
Description: TEAEs are defined as AEs which had onset on or after the start date and time of initial study medication administration. The SS consisted of all enrolled study participants who took at least 1 dose of the randomized treatment. Eligible participants who did not undergo any treatment of lacosamide but experienced an AE, are presented in a separate group "No Treatment".
Arm/Group | No Treatment | Active Comparator | Lacosamide
All-Cause Mortality (participants affected / at risk) | 0/3 | 0/12 | 1/14
Serious Adverse Events (participants affected / at risk) | 0/3 | 0/12 | 2/14
Other Adverse Events (participants affected / at risk) | 1/3 | 5/12 | 8/14
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | No Treatment (N=3) | Active Comparator (N=12) | Lacosamide (N=14)
Congenital central nervous system anomaly (Congenital, familial and genetic disorders) | 0 (0) | 0 (0) | 1 (1)
Cerebral infarction (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | No Treatment (N=3) | Active Comparator (N=12) | Lacosamide (N=14)
Eosinophilia (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 1 (1)
Right ventricular hypertrophy (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0)
Adrenal insufficiency (Endocrine disorders) | 0 (0) | 1 (1) | 1 (1)
Adrenal haemorrhage (Endocrine disorders) | 0 (0) | 0 (0) | 1 (1)
Diabetes insipidus (Endocrine disorders) | 0 (0) | 1 (1) | 0 (0)
Dry eye (Eye disorders) | 0 (0) | 0 (0) | 1 (1)
Retinal haemorrhage (Eye disorders) | 0 (0) | 1 (1) | 0 (0)
Vomiting (Gastrointestinal disorders) | 0 (0) | 1 (1) | 2 (2)
Constipation (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1)
Pain (General disorders) | 0 (0) | 1 (2) | 0 (0)
Pyrexia (General disorders) | 0 (0) | 1 (2) | 0 (0)
Cholestasis (Hepatobiliary disorders) | 0 (0) | 1 (1) | 0 (0)
Hyperbilirubinaemia neonatal (Hepatobiliary disorders) | 0 (0) | 0 (0) | 1 (1)
Infection (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
Neonatal infection (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Oral candidiasis (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
Feeding disorder neonatal (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 1 (1)
Hyponatraemia (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 0 (0)
Convulsion (Nervous system disorders) | 0 (0) | 0 (0) | 2 (2)
Poor sucking reflex (Nervous system disorders) | 0 (0) | 1 (2) | 0 (0)
Reflexes abnormal (Nervous system disorders) | 0 (0) | 1 (2) | 0 (0)
Cerebral ischaemia (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0)
Cerebrospinal fluid leakage (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0)
Depressed level of consciousness (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0)
Intracranial pressure increased (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0)
Lethargy (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1)
Hypercapnia (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1)
Pulmonary hypertension (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1)
Pulmonary oedema (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1)
Skin lesion (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (1)
Hypertension (Vascular disorders) | 0 (0) | 0 (0) | 1 (1)
Elevated Alanine Aminotransferase (Investigations) | 1 (1) | 0 (0) | 0 (0)

LIMITATIONS AND CAVEATS:
The study ended prematurely after agreed PIP modification; the termination was not linked to any safety issues/reasons.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of more than 60 days

DOCUMENTS (2):
  • Study Protocol (2022-02-11): https://cdn.clinicaltrials.gov/large-docs/45/NCT04519645/Prot_000.pdf
  • Statistical Analysis Plan (2023-05-04): https://cdn.clinicaltrials.gov/large-docs/45/NCT04519645/SAP_001.pdf